CLINICAL TRIAL: NCT06266494
Title: Prevention and Treatment of Frostbite Infection With Antimicrobial Pharmacokinetic Analysis
Acronym: Frostbite
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1349; CDMRP-DM220077 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-01-29; First posted 2024-02-20 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Frostbite
MeSH Terms: conditions — Frostbite | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Aim 1: Aloe Vera (Active Comparator): Aloe Vera will be applied topically to participant's frostbitten tissues twice daily.
  Interventions: Other: Aloe Vera
- Aim 1: Long-Acting Silver Dressings (Experimental): Long-Acting Silver dressings will be applied topically to participant's frostbitten tissues every 4 days.
  Interventions: Device: Long-Acting silver dressings
- Aim 2: Dalbavancin (Experimental): Participants will receive one 1500mg dose of Dalbavancin intravenously.
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Device: Long-Acting silver dressings — Mepilex Transfer Ag
  Arms: Aim 1: Long-Acting Silver Dressings
Other: Aloe Vera — Dermaid Aloe Vera
  Arms: Aim 1: Aloe Vera
Drug: Dalbavancin — 1500mg IV dose
  Arms: Aim 2: Dalbavancin

SUMMARY:
This study will compare the effectiveness of two different treatments for preventing infection from frostbite injuries. These two treatments are A) aloe vera and B) long-acting silver wound dressings. The investigators will also study the safety and effectiveness of Dalbavancin, an FDA approved antibiotic used for treating people who develop frostbite wound infections, as well as evaluate how frostbite damage to individuals' bodies may affect how fast their kidney clear drugs from their systems.

ELIGIBILITY:
Inclusion Criteria:

* All aims, aged ≥18 - < 99 years old admitted to UCH Burn Center with frostbite injury
* Aim 1: Admitted to UCH Burn Center with acute (within 4 days of cold exposure) frostbite injury
* Aim 2: Admitted to UCH Burn center with a clinically confirmed or suspected infected frostbite wound

Exclusion Criteria:

* Pregnant patients
* Prisoners
* Anticipated death within 48 hours of admission
* Inability to obtain consent from patient, legally authorized representative, or proxy
* Aim 1:Patients admitted five days and later from frostbite injury. Patients who have a clinical infection at baseline. Any patients that have a contra-indication for the use of either aloe (allergy), or silver (allergy).
* Aim 2: Any patients that have a contraindication for use of dalbavancin, including known history of hypersensitivity to dalbavancin, vancomycin, or other glycopeptide antibiotics. Patients with infections known to be caused by vancomycin-resistant Enterococcus; or those with Stage IV or V chronic kidney disease, or with cirrhosis (Childs-Pugh C); or those with anticipated death within 48 hours of infection.
* Aim 3: Anuria due to chronic kidney disease (CKD)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The number of positive microbial wound cultures on admission | Admission
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 4 | Hospital Day 4
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 8 | Hospital Day 8
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 12 | Hospital Day 12
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 16 | Hospital Day 16
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 20 | Hospital Day 20
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 24 | Hospital Day 24
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 28 | Hospital Day 28
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 32 | Hospital Day 32
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 36 | Hospital Day 36
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 40 | Hospital Day 40
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 44 | Hospital Day 44
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 48 | Hospital Day 48
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 52 | Hospital Day 52
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 56 | Hospital Day 56
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
The number of positive microbial wound cultures on hospital day 60 | Hospital Day 60
  Aerobic wound swabs will be taken from area of frostbite injury and analyzed by the (University of Colorado Hospital) UCH clinical laboratory. A positive culture indicates an organism was identified by the wound swab.
Number of gram positive cultures at admission | Admission
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 4 | Hospital Day 4
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 8 | Hospital Day 8
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 12 | Hospital Day 12
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 16 | Hospital Day 16
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 20 | Hospital Day 20
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 24 | Hospital Day 24
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 28 | Hospital Day 28
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 32 | Hospital Day 32
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 36 | Hospital Day 36
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 40 | Hospital Day 40
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 44 | Hospital Day 44
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 48 | Hospital Day 48
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 52 | Hospital Day 52
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 56 | Hospital Day 56
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Number of gram positive cultures on hospital day 60 | Hospital Day 60
  UCH clinical laboratory will identify cultures using MALDI-TOF MS (Matrix-Assisted Laser Desorption - Ionisation-Time of Flight Mass Spectrometry).
Change in serum concentration of dalbavancin in plasma (mcg/ml) over time | 1, 4, 12 hours, and 1,2,3,4,6,8,10,13,16 (or date of discharge if earlier) days post dalbavancin infusion
Dalbavancin concentrations in subcutaneous tissue | Up to 12 weeks
  Dalbavancin concentration measured in frostbitten subcutaneous tissue by mcg/g
Change in presence of Augmented Renal Clearance | Baseline, Up to 12 weeks
  Creatinine clearance will be calculated from a 12-hour urine collection, with the definition of Augmented Renal Clearance as: CrCl > 130mL/min.

CONTACTS AND LOCATIONS:
Overall Officials: Arek Wiktor, MD, Principal Investigator — University of Colorado Anschtuz
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undetermined at this time

REFERENCES:
- [Background] Mueller SW, Blass B, Molina KC, Gibson C, Krsak M, Kohler AD, Deeter L, Stalilonis J, Wiktor AJ. Augmented Renal Function in Burn Patients: Occurrence and Discordance With Commonly Used Methods to Assess Renal Function. J Burn Care Res. 2023 Nov 2;44(6):1298-1303. doi: 10.1093/jbcr/irad107. PMID 37450897
- [Background] Carmichael H, Michel S, Smith TM, Duffy PS, Wiktor AJ, Lambert Wagner A. Remote Delivery of Thrombolytics Prior to Transfer to a Regional Burn Center for Tissue Salvage in Frostbite: A Single-center Experience of 199 Patients. J Burn Care Res. 2022 Jan 5;43(1):54-60. doi: 10.1093/jbcr/irab041. PMID 33657205
- [Background] Torian SC, Wiktor AJ, Roper SE, Laramie KE, Miller MA, Mueller SW. Burn Injury and Augmented Renal Clearance: A Case for Optimized Piperacillin-Tazobactam Dosing. J Burn Care Res. 2023 Jan 5;44(1):203-206. doi: 10.1093/jbcr/irac138. PMID 36173707
- [Background] Barletta JF, Mangram AJ, Byrne M, Sucher JF, Hollingworth AK, Ali-Osman FR, Shirah GR, Haley M, Dzandu JK. Identifying augmented renal clearance in trauma patients: Validation of the Augmented Renal Clearance in Trauma Intensive Care scoring system. J Trauma Acute Care Surg. 2017 Apr;82(4):665-671. doi: 10.1097/TA.0000000000001387. PMID 28129261
- [Background] Udy AA, Jarrett P, Stuart J, Lassig-Smith M, Starr T, Dunlop R, Wallis SC, Roberts JA, Lipman J. Determining the mechanisms underlying augmented renal drug clearance in the critically ill: use of exogenous marker compounds. Crit Care. 2014 Nov 29;18(6):657. doi: 10.1186/s13054-014-0657-z. PMID 25432141
- [Background] Cook AM, Hatton-Kolpek J. Augmented Renal Clearance. Pharmacotherapy. 2019 Mar;39(3):346-354. doi: 10.1002/phar.2231. Epub 2019 Mar 11. PMID 30723936
- [Background] Dunne MW, Puttagunta S, Giordano P, Krievins D, Zelasky M, Baldassarre J. A Randomized Clinical Trial of Single-Dose Versus Weekly Dalbavancin for Treatment of Acute Bacterial Skin and Skin Structure Infection. Clin Infect Dis. 2016 Mar 1;62(5):545-51. doi: 10.1093/cid/civ982. Epub 2015 Nov 26. PMID 26611777
- [Background] Carrothers TJ, Chittenden JT, Critchley I. Dalbavancin Population Pharmacokinetic Modeling and Target Attainment Analysis. Clin Pharmacol Drug Dev. 2020 Jan;9(1):21-31. doi: 10.1002/cpdd.695. Epub 2019 May 14. PMID 31087630
- [Background] Mangum LC, Garcia GR, Akers KS, Wenke JC. Duration of extremity tourniquet application profoundly impacts soft-tissue antibiotic exposure in a rat model of ischemia-reperfusion injury. Injury. 2019 Dec;50(12):2203-2214. doi: 10.1016/j.injury.2019.09.025. Epub 2019 Sep 20. PMID 31591007
- [Background] Kam PC, Kavanagh R, Yoong FF. The arterial tourniquet: pathophysiological consequences and anaesthetic implications. Anaesthesia. 2001 Jun;56(6):534-45. doi: 10.1046/j.1365-2044.2001.01982.x. PMID 11412159
- [Background] Dunne MW, Puttagunta S, Sprenger CR, Rubino C, Van Wart S, Baldassarre J. Extended-duration dosing and distribution of dalbavancin into bone and articular tissue. Antimicrob Agents Chemother. 2015 Apr;59(4):1849-55. doi: 10.1128/AAC.04550-14. Epub 2015 Jan 5. PMID 25561338
- [Background] Nicolau DP, Sun HK, Seltzer E, Buckwalter M, Dowell JA. Pharmacokinetics of dalbavancin in plasma and skin blister fluid. J Antimicrob Chemother. 2007 Sep;60(3):681-4. doi: 10.1093/jac/dkm263. Epub 2007 Jul 12. PMID 17631507
- [Background] Morrisette T, Miller MA, Montague BT, Barber GR, McQueen RB, Krsak M. On- and off-label utilization of dalbavancin and oritavancin for Gram-positive infections. J Antimicrob Chemother. 2019 Aug 1;74(8):2405-2416. doi: 10.1093/jac/dkz162. PMID 31322694
- [Background] Molina KC, Lunowa C, Lebin M, Segerstrom Nunez A, Azimi SF, Krsak M, Mueller SW, Miller MA. Comparison of Sequential Dalbavancin With Standard-of-Care Treatment for Staphylococcus aureus Bloodstream Infections. Open Forum Infect Dis. 2022 Jul 14;9(7):ofac335. doi: 10.1093/ofid/ofac335. eCollection 2022 Jul. PMID 35899276
- [Background] Cain AR, Bremmer DN, Carr DR, Buchanan C, Jacobs M, Walsh TL, Moffa MA, Shively NR, Trienski TL. Effectiveness of Dalbavancin Compared With Standard of Care for the Treatment of Osteomyelitis: A Real-world Analysis. Open Forum Infect Dis. 2021 Dec 18;9(2):ofab589. doi: 10.1093/ofid/ofab589. eCollection 2022 Feb. PMID 35071682
- [Background] Rappo U, Puttagunta S, Shevchenko V, Shevchenko A, Jandourek A, Gonzalez PL, Suen A, Mas Casullo V, Melnick D, Miceli R, Kovacevic M, De Bock G, Dunne MW. Dalbavancin for the Treatment of Osteomyelitis in Adult Patients: A Randomized Clinical Trial of Efficacy and Safety. Open Forum Infect Dis. 2018 Dec 10;6(1):ofy331. doi: 10.1093/ofid/ofy331. eCollection 2019 Jan. PMID 30648126
- [Background] Boucher HW, Wilcox M, Talbot GH, Puttagunta S, Das AF, Dunne MW. Once-weekly dalbavancin versus daily conventional therapy for skin infection. N Engl J Med. 2014 Jun 5;370(23):2169-79. doi: 10.1056/NEJMoa1310480. PMID 24897082
- [Background] Jones RN, Fritsche TR, Sader HS, Goldstein BP. Antimicrobial spectrum and potency of dalbavancin tested against clinical isolates from Europe and North America (2003): initial results from an international surveillance protocol. J Chemother. 2005 Dec;17(6):593-600. doi: 10.1179/joc.2005.17.6.593. PMID 16433188
- [Background] Molina KC, Miller MA, Mueller SW, Van Matre ET, Krsak M, Kiser TH. Clinical Pharmacokinetics and Pharmacodynamics of Dalbavancin. Clin Pharmacokinet. 2022 Mar;61(3):363-374. doi: 10.1007/s40262-021-01088-w. Epub 2021 Dec 21. PMID 34931283
- [Background] Sader HS, Castanheira M, Huband MD, Shortridge D, Carvalhaes CG, Mendes RM. Antimicrobial activity of dalbavancin against Gram-positive bacteria isolated from patients hospitalized with bloodstream infection in United States and European medical centers (2018-2020). Eur J Clin Microbiol Infect Dis. 2022 May;41(5):867-873. doi: 10.1007/s10096-022-04437-0. Epub 2022 Mar 30. PMID 35355158
- [Background] Goldstein EJ, Citron DM, Warren YA, Tyrrell KL, Merriam CV, Fernandez HT. In vitro activities of dalbavancin and 12 other agents against 329 aerobic and anaerobic gram-positive isolates recovered from diabetic foot infections. Antimicrob Agents Chemother. 2006 Aug;50(8):2875-9. doi: 10.1128/AAC.00286-06. PMID 16870792
- [Background] Madry R, Struzyna J, Stachura-Kulach A, Drozdz L, Bugaj M. Effectiveness of Suprathel(R) application in partial thickness burns, frostbites and Lyell syndrome treatment. Pol Przegl Chir. 2011 Oct;83(10):541-8. doi: 10.2478/v10035-011-0086-5. PMID 22189281
- [Background] Heil K, Thomas R, Robertson G, Porter A, Milner R, Wood A. Freezing and non-freezing cold weather injuries: a systematic review. Br Med Bull. 2016 Mar;117(1):79-93. doi: 10.1093/bmb/ldw001. Epub 2016 Feb 12. PMID 26872856
- [Background] Gonzaga T, Jenabzadeh K, Anderson CP, Mohr WJ, Endorf FW, Ahrenholz DH. Use of Intra-arterial Thrombolytic Therapy for Acute Treatment of Frostbite in 62 Patients with Review of Thrombolytic Therapy in Frostbite. J Burn Care Res. 2016 Jul-Aug;37(4):e323-34. doi: 10.1097/BCR.0000000000000245. PMID 25950290
- [Background] Goertz O, Hirsch T, Buschhaus B, Daigeler A, Vogelpohl J, Langer S, Steinau HU, Ring A. Intravital pathophysiologic comparison of frostbite and burn injury in a murine model. J Surg Res. 2011 May 15;167(2):e395-401. doi: 10.1016/j.jss.2011.01.034. Epub 2011 Feb 18. PMID 21392800
- [Background] Cauchy E, Cheguillaume B, Chetaille E. A controlled trial of a prostacyclin and rt-PA in the treatment of severe frostbite. N Engl J Med. 2011 Jan 13;364(2):189-90. doi: 10.1056/NEJMc1000538. No abstract available. PMID 21226604
- [Background] Imray C, Grieve A, Dhillon S; Caudwell Xtreme Everest Research Group. Cold damage to the extremities: frostbite and non-freezing cold injuries. Postgrad Med J. 2009 Sep;85(1007):481-8. doi: 10.1136/pgmj.2008.068635. PMID 19734516
- [Background] Woodmansey EJ, Roberts CD. Appropriate use of dressings containing nanocrystalline silver to support antimicrobial stewardship in wounds. Int Wound J. 2018 Dec;15(6):1025-1032. doi: 10.1111/iwj.12969. Epub 2018 Aug 17. PMID 30117675
- [Background] Silverstein P, Heimbach D, Meites H, Latenser B, Mozingo D, Mullins F, Garner W, Turkowski J, Shupp J, Glat P, Purdue G. An open, parallel, randomized, comparative, multicenter study to evaluate the cost-effectiveness, performance, tolerance, and safety of a silver-containing soft silicone foam dressing (intervention) vs silver sulfadiazine cream. J Burn Care Res. 2011 Nov-Dec;32(6):617-26. doi: 10.1097/BCR.0b013e318236fe31. PMID 21979855
- [Background] Norman G, Christie J, Liu Z, Westby MJ, Jefferies JM, Hudson T, Edwards J, Mohapatra DP, Hassan IA, Dumville JC. Antiseptics for burns. Cochrane Database Syst Rev. 2017 Jul 12;7(7):CD011821. doi: 10.1002/14651858.CD011821.pub2. PMID 28700086
- [Background] Dat AD, Poon F, Pham KB, Doust J. Aloe vera for treating acute and chronic wounds. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008762. doi: 10.1002/14651858.CD008762.pub2. PMID 22336851
- [Background] Miller MB, Koltai PJ. Treatment of experimental frostbite with pentoxifylline and aloe vera cream. Arch Otolaryngol Head Neck Surg. 1995 Jun;121(6):678-80. doi: 10.1001/archotol.1995.01890060076015. PMID 7772322
- [Background] Klein AD, Penneys NS. Aloe vera. J Am Acad Dermatol. 1988 Apr;18(4 Pt 1):714-20. doi: 10.1016/s0190-9622(88)70095-x. PMID 3286692
- [Background] Heggers JP, Robson MC, Manavalen K, Weingarten MD, Carethers JM, Boertman JA, Smith DJ Jr, Sachs RJ. Experimental and clinical observations on frostbite. Ann Emerg Med. 1987 Sep;16(9):1056-62. doi: 10.1016/s0196-0644(87)80758-8. PMID 3631670
- [Background] Khaira HS, Coddington T, Drew A, Roberts PN, Imray CH. Patellar tendon bearing orthosis--application as adjunctive treatment in healing of lower-limb tissue loss. Eur J Vasc Endovasc Surg. 1998 Dec;16(6):485-8. doi: 10.1016/s1078-5884(98)80238-4. PMID 9894487
- [Background] Imray CH, Oakley EH. Cold still kills: cold-related illnesses in military practice freezing and non-freezing cold injury. J R Army Med Corps. 2005 Dec;151(4):218-22. doi: 10.1136/jramc-151-04-02. No abstract available. PMID 16548337
- [Background] Cauchy E, Chetaille E, Marchand V, Marsigny B. Retrospective study of 70 cases of severe frostbite lesions: a proposed new classification scheme. Wilderness Environ Med. 2001 Winter;12(4):248-55. doi: 10.1580/1080-6032(2001)012[0248:rsocos]2.0.co;2. PMID 11769921
- [Background] Cauchy E, Marsigny B, Allamel G, Verhellen R, Chetaille E. The value of technetium 99 scintigraphy in the prognosis of amputation in severe frostbite injuries of the extremities: A retrospective study of 92 severe frostbite injuries. J Hand Surg Am. 2000 Sep;25(5):969-78. doi: 10.1053/jhsu.2000.16357. PMID 11040315
- [Background] Handford C, Thomas O, Imray CHE. Frostbite. Emerg Med Clin North Am. 2017 May;35(2):281-299. doi: 10.1016/j.emc.2016.12.006. PMID 28411928
- [Background] Zaramo TZ, Green JK, Janis JE. Practical Review of the Current Management of Frostbite Injuries. Plast Reconstr Surg Glob Open. 2022 Oct 24;10(10):e4618. doi: 10.1097/GOX.0000000000004618. eCollection 2022 Oct. PMID 36299821
- [Background] Bruen KJ, Ballard JR, Morris SE, Cochran A, Edelman LS, Saffle JR. Reduction of the incidence of amputation in frostbite injury with thrombolytic therapy. Arch Surg. 2007 Jun;142(6):546-51; discussion 551-3. doi: 10.1001/archsurg.142.6.546. PMID 17576891
- [Background] Bennett BL, Holcomb JB. Battlefield Trauma-Induced Hypothermia: Transitioning the Preferred Method of Casualty Rewarming. Wilderness Environ Med. 2017 Jun;28(2S):S82-S89. doi: 10.1016/j.wem.2017.03.010. Epub 2017 May 5. PMID 28483389
- [Background] DeGroot DW, Rappole CA, McHenry P, Englert RM. Seasonal Trends for Environmental Illness Incidence in the U.S. Army. Mil Med. 2022 May 3;187(5-6):e672-e677. doi: 10.1093/milmed/usab072. PMID 33605408